CLINICAL TRIAL: NCT05003219
Title: Long Term Clinical Outcome of Single Open Door Laminoplasty With Preservation of Unilateral Muscular Ligament Complex
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2021009
Record Dates: First submitted 2021-07-01; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-06

CONDITIONS: Cervical Myelopathy
Keywords: Open Door Laminoplasty; Preservation of Unilateral Muscular Ligament Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERAS group: patients received posterior cervical open-door laminoplasty under ERAS mode
- Conventional group: patients received posterior cervical open-door laminoplasty under routine perioperative management mode

SUMMARY:
To collect and measure the preoperative and postoperative clinical data of the patients undergoing single open-door expansive laminoplasty with preservation of musclar ligament complex through posterior cervical approach in our hospital and summarize the long-term clinical effect and postoperative imaging changes and analyze the long-term clinical effect of this operation

DETAILED DESCRIPTION:
Objective: To collect and measure the preoperative and postoperative clinical data of the patients undergoing single open-door expansive laminoplasty with preservation of musclar ligament complex through posterior cervical approach in our hospital. To summarize the long-term clinical effect and postoperative imaging changes and to analyze the long-term clinical effect of this operation on cervical spondylosis. To provide scientific basis for clinical work and theoretical research in the future.

This study was a retrospective study, and the medical records of posterior cervical open-door expansive laminoplasty with musclar ligament complex preservation in the orthopedics department of our hospital from 2006 to 2017 were collected, and the patients with complete diagnosis and treatment data were selected for analysis and research.The preoperative and postoperative changes of the patients were studied by combining the patient's case and imaging examination (MR, CT, X plain film) and other diagnosis and treatment data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70, gender unlimited;
2. The patient was diagnosed with cervical spondylosis and met the indications of posterior cervical laminoplasty;
3. Basis of serious diseases of heart, brain, lung, kidney or other important organs, preoperative ASA score I-II;
4. Agree to participate in the study and sign the informed consent；

Exclusion Criteria:

1. Preoperative ASA score ≥III;
2. One-stage combined anterior and posterior surgery of cervical spine;
3. Correction of cervical deformity;
4. Patients with gastric emptied disorders (such as gastroesophageal reflux, chronic history of aspiration, delayed gastric emptied), complete obstruction of the digestive tract, and inability to use enteral preparations;
5. Patients with high risk conditions, such as severe cardio-renal insufficiency, affecting the safety evaluation of the trial;
6. People with mental disorders, alcohol dependence or drug abuse history;
7. women in the period of lactation and pregnancy;
8. People with allergic constitution or previous allergies to a variety of drugs;
9. Other researchers consider it inappropriate to participate in this study

Age Groups: Child, Adult, Older Adult
Study Population: Between August 2020 and December 2021, patients receiving conventional cervical posterior open-door laminoplasty due to cervical myelopathy or ossification of the posterior longitudinal ligament of the cervical spine
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
mJOA | 2 years after operation
  Modified Japanese Orthopaedic Association score
neck and shoulder VAS | 2 years after operation
  neck and shoulder visual analogue score
NDI | 2 years after operation
  neck disability index
AS | 2 years after operation
  axial syndrome
C5 palsy | 2 years after operation
  C5 palsy after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No